CLINICAL TRIAL: NCT00880386
Title: A Pilot Project to Determine the Effect of Losartan (Cozaar) on Radiation-Induced Pulmonary Fibrosis in Patients With Non-Small Cell Lung Cancer
Brief Title: Losartan in Treating Pulmonary Fibrosis in Patients With Stage I, II, or III Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study concept was not approved by NCI. Study was never activated. No enrollment
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCUSF 0208; SCUSF-PILOT-0208 (Other: SunCoast CCOP Research Base); HLMCC-PILOT-0208 (Other: H. Lee Moffitt Cancer Center Research Base)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Dyspnea; Lung Cancer; Pulmonary Complications; Radiation Fibrosis
Keywords: dyspnea; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; pulmonary complications; radiation fibrosis
MeSH Terms: conditions — Dyspnea; Lung Neoplasms; Radiation Fibrosis Syndrome; Carcinoma, Non-Small-Cell Lung | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Losartan Group (Experimental): 50 mg Losartan tablet taken daily for 24 weeks
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — 50 mg Losartan will be taken daily by subjects for 24 weeks
  Other Names: Cozaar; losartan potassium

SUMMARY:
RATIONALE: Losartan potassium may be effective in treating pulmonary fibrosis caused by radiation therapy in patients with non-small cell lung cancer.

PURPOSE: This clinical trial is studying losartan to see how well it works in treating pulmonary fibrosis caused by radiation therapy in patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effects of losartan potassium on the disease progression in patients with stage I-III non-small cell lung cancer and radiation-induced pulmonary fibrosis.
* To determine the feasibility of losartan potassium as a possible treatment for radiation-induced pulmonary fibrosis.

Secondary

* The evaluate the effects of losartan potassium on the degree of dyspnea, and lung function (FEV_1 and FVC) in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral losartan potassium once daily for 6 months in the absence of disease progression or unacceptable toxicity.

Patients undergo assessment of pulmonary function (e.g., gas movement, lung capacity, and diffusion of gases) by spirometry and dyspnea by the Visual Analog Scale (VAS) at baseline and at weeks 12 and 24.

ELIGIBILITY:
INCLUSION CRITERIA:

* At least 18 years of age or older
* Diagnosed with non-small cell lung cancer stage I, II, IIIa, or IIIb
* Diagnosis of radiation-induced pulmonary fibrosis (as defined by National Cancer Institute's Common Terminology Criteria for Adverse Events [CTCAE] V3.0 Grade I to Grade III) and within 2 years of the last radiation therapy treatment

EXCLUSION CRITERIA:

* Patients with a pneumonectomy
* Allergy or allergic reaction to Losartan or any other angiotensin II receptor blocker
* Use of an angiotensin II receptor blocker currently or within 6 months of study entry which include: losartan, valsartan, irbesartan, candesartan, cilexetil, eprosartan mesylate, and telmisartan
* Bilateral renal artery stenosis, hereditary or idiopathic angioedema, or uncontrolled hypotension
* Patients taking lithium
* Currently smoking or smoked within 6 months of study entry
* Pregnant, intending to become pregnant or breastfeeding
* Baseline systolic blood pressure < 100 mmHg
* History of lung transplant
* History of kidney failure or liver disease
* Inability to attend clinic visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in carbon monoxide diffusing capacity (DLCO) at 6 months | 6 months

SECONDARY OUTCOMES:
Feasibility of losartan potassium as treatment for radiation-induced pulmonary fibrosis | 6 months
Pulmonary function measurements of FEV1 and FVC and dyspnea score at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Couluris, DO, Principal Investigator — University of South Florida